CLINICAL TRIAL: NCT04027751
Title: The Efficacy and Safety of Tropisetron in Preventing Emergence Delirium: A Randomized Controlled Trial
Brief Title: The Efficacy and Safety of Tropisetron in Preventing Emergence Delirium
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Chao Yang Hospital (Other)
Responsible Party: Principal Investigator, Anshi Wu, Head of Anesthesiology, Beijing Chao Yang Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 04719372
Record Dates: First submitted 2019-07-16; First posted 2019-07-22 (Actual); Last update posted 2020-03-11 (Actual); Status verified 2020-03

CONDITIONS: Emergence Delirium; Postoperative Delirium
Keywords: tropisetron; emergence delirium; postoperative delirium
MeSH Terms: conditions — Emergence Delirium | interventions — Tropisetron

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tropisetron (Experimental): Patients allocated to this arm will receive single dose of intravenous Tropisetron (5mg) before anesthesia induction.
  Interventions: Drug: Tropisetron
- Placebo (Placebo Comparator): Patients allocated to this arm will receive an identical volume of saline solution before anesthesia induction.
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Tropisetron — Investigators administrated intravenously Tropisetron 5mg before anesthesia induction
  Arms: Tropisetron
Drug: Placebos — Investigators administrated intravenously 0.9% saline solution as a placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the efficacy and safety of Tropisetron in preventing emergence delirium.

DETAILED DESCRIPTION:
Delirium is a common complication during postoperative period, especially in elderly patients. The presence of postoperative delirium is independently associated with poor recovery, increased length of hospital stay, the development of long-term cognitive decline and increased mortality.

Tropisetron is a 5-HT3A receptor antagonist and is widely used to treat postoperative nausea and vomiting. Previous studies found that tropisetron has positive effect on cognitive function. This study aims to access the efficacy and safety of tropisetron in preventing emergence delirium.

To explore the results differences amongst different patients, subgroup analysis will be conducted according to: a. Age (older than 65 years versus 65 years or younger); b. Surgery type (major surgery versus minor surgery); c. Preoperative MoCA scores (>26 versus 18-26 versus 10-17).

ELIGIBILITY:
Inclusion Criteria:

1. Written consent given
2. Scheduled to undergo elective non-cardiac surgeries under general anesthesia
3. ASA Physical Score I-III

Exclusion Criteria:

1. Patients with a history of neurological disease, such as Alzheimer disease.
2. Patients with a history of psychiatric disease
3. Patients with a medication history of antipsychotic drugs over the last 30 days prior to enrollment.
4. Unable to complete neuropsychological testing including patients with severe visual or hearing impairment.
5. the Montreal Cognitive Assessment (MoCA) scores below 10
6. Patients who have severe intraoperative adverse events, such as cardiac arrest.
7. Patients with contraindication of tropisetron.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1508 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-03-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of emergence delirium | Until the end of post-anesthesia care unit stay, assessed up to 1 hour
  Screening of the patients regarding an emergence delirium by The Confusion Assessment Method for The Intensive Care Unit (CAM-ICU). CAM-ICU is assessed at three different points of time:
  1. 15min after excubation
  2. 30min after excubation
  3. At discharge from post-anesthesia care unit (PACU)

SECONDARY OUTCOMES:
Incidence of postoperative delirium | Within 3 days after surgery
  Screening of the patients regarding a postoperative delirium by The Confusion Assessment Method for The Intensive Care Unit (CAM-ICU)
Incidence of postoperative nausea and vomiting | Within 3 days after surgery
Postoperative Pain | Within 3 days after surgery
  Visual Analogue Scale will be used to assess postoperative pain of patients. Numerical rating scale ranging from 0 to 10, where 0 indicates no pain and 10 indicates the worst pain.
Length of Hospital stay | From the date of admission until discharged from hospital, up to 30 days
Adverse events | Within 3 days after surgery
  Other adverse events within 3 days after surgery were noted

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Chaoyang Hospital, Capital Medical University, Beijing, China

REFERENCES:
- [Derived] Huang X, Wu D, Wu AS, Wei CW, Gao JD. The Association of Insomnia with Depression and Anxiety Symptoms in Patients Undergoing Noncardiac Surgery. Neuropsychiatr Dis Treat. 2021 Mar 25;17:915-924. doi: 10.2147/NDT.S296986. eCollection 2021. PMID 33790560
- [Derived] Sun Y, Lin D, Wang J, Geng M, Xue M, Lang Y, Cui L, Hao Y, Mu S, Wu D, Liang L, Wu A; Tropisetron and Delirium Group. Effect of Tropisetron on Prevention of Emergence Delirium in Patients After Noncardiac Surgery: A Trial Protocol. JAMA Netw Open. 2020 Oct 1;3(10):e2013443. doi: 10.1001/jamanetworkopen.2020.13443. PMID 33052400